CLINICAL TRIAL: NCT00425646
Title: A Phase II Study Evaluating a Maintenance Strategy of Gleevce® (Imatinib Mesylate) and Bevacizumab in Patients With Advanced, Non-squamous, Non-small Cell Lung Cancer, Following Completion of First-line Chemotherapy With Bevacizumab
Brief Title: Imatinib Mesylate and Bevacizumab After First-Line Chemotherapy and Bevacizumab in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Laurie Carr, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Masking: None | Purpose: Treatment
Other Study IDs: 6351; UWCC-6351; UWCC-06-3622-H/B; NOVARTIS-UWCC-6351; CDR0000526130 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Imatinib Mesylate

INTERVENTIONS:
Biological: bevacizumab
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Imatinib mesylate and bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving imatinib mesylate together with bevacizumab as maintenance therapy may stop non-small cell lung cancer from growing or coming back.

PURPOSE: This phase II trial is studying how well giving imatinib mesylate together with bevacizumab after first-line chemotherapy and bevacizumab works in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical efficacy of maintenance therapy comprising imatinib mesylate and bevacizumab after completion of first-line, platinum-based chemotherapy and bevacizumab, in terms of progression-free survival, in patients with stage IIIB or IV non-small cell lung cancer.

Secondary

* Assess the safety profile of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral imatinib mesylate twice daily on days 1-21 and bevacizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIB (by pleural effusion only) or stage IV disease
  * No predominately squamous cell carcinoma

    * Mixed tumors will be categorized by predominant cell type
* Must have completed 4 courses of platinum-based, doublet chemotherapy and bevacizumab*, has no disease progression, and meets the following criteria:

  * Platinum agent may have included carboplatin or cisplatin
  * Second agent may have included paclitaxel, docetaxel, gemcitabine hydrochloride, vinorelbine ditartrate, or pemetrexed disodium
  * A change in the platinum doublet is acceptable provided the following are true:

    * Basis for change was toxicity rather than disease progression
    * Total number of courses of any platinum doublet plus bevacizumab was 4
  * At least 3 of 4 courses must have included bevacizumab NOTE: *Patients age 70 and over may have completed 4 courses of single-agent chemotherapy plus bevacizumab; single agent chemotherapy may have included paclitaxel, docetaxel, gemcitabine hydrochloride, vinorelbine ditartrate, or pemetrexed disodium
* No brain metastases by brain MRI or head CT scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Absolute neutrophil count ≥ 1500/mm³
* Platelet count ≥ 100,000/mm³
* INR ≤ 1.5 times ULN
* Urine protein:creatinine ratio ≤ 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* No history of gross hemoptysis (defined as > ½ teaspoon of bright red blood)
* No inadequately controlled hypertension (defined as blood pressure > 150/100 mm Hg on antihypertensive medications)
* No significant traumatic injury within the past 28 days
* No condition requiring continuous administration of systemic corticosteroids
* No medical condition that would preclude study treatment
* No medical comorbidities, including any of the following:

  * Unstable angina
  * Congestive heart failure ≥ grade 2
  * Myocardial infarction within the past 6 months
  * Stroke within the past 6 months
  * Peripheral vascular disease ≥ grade 2 within the past 6 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy in the metastatic setting, except for 4 courses of platinum-based, doublet chemotherapy plus bevacizumab in the first-line setting

  * Prior adjuvant, neoadjuvant, or combined modality chemoradiation for localized non-small cell lung cancer allowed provided ≥ 6 months elapsed before metastatic recurrence
* At least 28 days since prior major surgical procedure
* No prior antiangiogenic drug, including AMG 706, CP-547, 632, vatalanib, AZD2171, thalidomide, sorafenib tosylate, or sunitinib malate
* No other concurrent investigational drugs
* No concurrent grapefruit juice or products containing grapefruit
* No other concurrent anticancer agents, including chemotherapy and biological agents
* No concurrent major surgical procedure
* No concurrent therapeutic coagulation comprising warfarin, heparin, or low molecular weight heparin

  * Low-dose warfarin (e.g., 1 mg/day) for prophylaxis of central venous catheter thrombosis allowed
* No chronic daily acetylsalicylic acid (> 325 mg/day) or other full-dose nonsteroidal anti-inflammatory drug with antiplatelet activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Toxicity rate, defined as percentage of patients experiencing a grade 3 or greater adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Carr, MD, Study Chair — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States